CLINICAL TRIAL: NCT06160882
Title: Evaluation of Powered Prosthesis for Use With Transfemoral Osseointegration Recipients
Brief Title: Powered Prosthesis for Use With TF Osseointegration Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern University (Other); Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Levi Hargrove, Director and Scientific Chair, Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00215805
Record Dates: First submitted 2023-08-29; First posted 2023-12-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Amputation
Keywords: Transfemoral Amputation
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The primary endpoint will be to evaluate the functional, biomechanical, metabolic outcomes, and user satisfaction while using a powered prosthesis suspended by an OI interface compared to their prescribed traditional socket
  The secondary endpoint will be to determine changes in EMG signal quality and neural information resulting from OI and TMR as compared to an instrumented socket for control of a powered leg prosthesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluation of Powered Prosthesis for use with Transfemoral Osseointegration Recipients (Other): Perform Osseointegration (OI)Surgery and Targeted Muscle Reinnervation (TMR) and evaluate powered prosthesis training and use. The participant will complete non-weightbearing neural control tasks along with functional, biomechanical, metabolic and qualitative patient-reported outcome measures using the OI interface and the powered leg prosthesis.
  Interventions: Other: Powered Prosthesis Training and EMG data collection; Procedure: Perform Osseointegration (OI) surgery and Targeted Muscle Reinnervation (TMR)

INTERVENTIONS:
Other: Powered Prosthesis Training and EMG data collection — Participants are fit for a custom instrumented socket for collection of surface EMG signals and use with the powered lower limb prosthesis.
  EMG control sites will be located using clinical best practices. Once socket fit is completed, the prosthetist will attach and align the powered prosthesis. The participant will be instructed to walk with the powered prosthesis for level ground walking, incline walking, stair climbing and non-weight bearing independence control activities. A non-weight bearing independent control system will be configured. These data are used to train a pattern recognition control system which can control the leg knee and ankle joints respectively, either in a virtual environment or with the physical prosthesis The participants will complete functional, biomechanical, metabolic, and patient reported outcome measures.
Procedure: Perform Osseointegration (OI) surgery and Targeted Muscle Reinnervation (TMR) — Participants will undergo OI Surgery 1 +TMR and recovery. Following recovery, participants will receive OI surgery 2 where the abutment is connected to the fixture with in the femur. Participants will receive standard post-surgical care and participate in the OPRA rehab program through the Shirley Ryan AbilityLab. The participant uses their clinically prescribed prosthetic knee unit for training in the OPRA rehab program.
  Post-Surgery Fitting and Powered Leg Prosthesis Training: EMG signals are measured using a custom fit electrode band on the residual limb that is tethered to the prosthesis. Participants are fit with the powered prosthesis using their OI interface and trained on its use. The participant will complete non-weight-bearing neural control tasks as done prior to surgery. The participants will complete functional, biomechanical, metabolic, and patient-reported outcome measures using the OI interface and the powered leg prosthesis.

SUMMARY:
The purpose of this study is to evaluate functional mobility, control, and user satisfaction from persons who have an amputation above the knee and have received osseo-integration (OI) and targeted muscle reinnervation (TMR) surgery, while walking with a powered knee and ankle prosthesis.

DETAILED DESCRIPTION:
The objective of this study is to evaluate functional mobility, non-weight-bearing neural control, and user satisfaction from individuals with unilateral transfemoral amputation who have received osseo-integration (OI) and targeted muscle reinnervation (TMR), while ambulating with a fully powered prosthesis.

The hypothesis is that OI will show perceived benefits for participants including: 1) lower perceived weight of the prosthesis due to the more secure OI interface over a traditional socket, 2) decreased energy expenditure during ambulation and transitions, and 3) electromyographic (EMG) signals will be higher quality and more robust than signals measured from within a socket, potentially allowing for improved pattern recognition driven prostheses in future device design and studies.

Prior to surgical intervention, amputee participants will visit the lab up to 3 times for socket fitting, and at most 7 times to practice using the powered prosthesis and collect experimental data. There is no time limitation between sessions and each session will last a maximum of 4 hours.

Aim 1: Pre-Surgery Fitting and Powered Leg Prosthesis Training:

Participants will be fit for a custom instrumented socket that allows for collection of surface EMG signals and for use with the powered lower limb prosthesis. The socket that is fabricated is solely for the purpose of this study, will be used only in the research lab. The participant will continue to use their clinically prescribed socket and prosthesis when not attending study visits. EMG control sites over the semitendinosus, biceps femoris, tensor fasciae latae, rectus femoris, vastus lateralis, and adductor magnus will be located using clinical best practices. Once socket fit is completed, the prosthetist will attach and align the powered prosthesis. The participant will be instructed to walk with the powered prosthesis for level ground walking, incline walking, stair climbing and non-weight bearing independence control activities. The walkway, ramps and stairs are equipped with handrails and the amputee with be wearing either an overhead harness or gait belt for safety. Additionally, a non-weight bearing independent control system will be configured. The participant will be instructed to attempt to move their 'phantom' limb through knee flexion/extension and ankle plantarflexion/dorsiflexion range movements while EMG data are collected. These data are used to train a pattern recognition control system which can control the leg knee and ankle joints respectively, either in a virtual environment or with the physical prosthesis. The participants will then complete functional, biomechanical, metabolic, and qualitative patient reported outcome measures using the instrumented socket and the powered leg prosthesis. The investigator will use an extensive list of standard clinical assessments and participant-reported measures that assess physical function, mobility, balance, fall risk, quality of life, and metabolic expenditure.

OI TMR surgery 1 and recovery: participants will undergo the first osseointegration (OI) and targeted muscle reinnervation (TMR) surgery at Northwestern Memorial Hospital.

OI surgery 2 and recovery: Participants will undergo the second OI surgery where the abutment will be connected to the fixture with in the femur. The participant will again be monitored for full recovery (typically 4-6 weeks). No outcome measures or assessments will be performed prior to 12 weeks' post-surgery

Aim 2: Post-Surgery Fitting and Powered Leg Prosthesis Training:

After osseointegration and TMR surgery and recovery, the study participant no longer requires a standard prosthetic socket. EMG signals can now be measured using a custom fit electrode band on the residual limb that is tethered to the prosthesis. Participants will be fit with the powered prosthesis using their OI interface and trained on its use. Participants will receive instruction on use of the powered prosthesis, now attached via their OI interface with the electrode band. The participants will walk under the supervision of a clinician while device parameters are configured as prior to OI/TMR surgery. The participant will progress to walking over slopes, perform stairclimbing with a reciprocal gait and sit to and from standing transitions. The clinician will provide verbal instruction and cues on how to best make use of the power and how to safely perform all activities. The investigators will repeat the same measures as previously performed to evaluate the functional, metabolic, and biomechanical benefits conferred by OI over a traditional socket when using a powered leg device. At the end of each visit, the study participant will return to their clinically prescribed prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower limb amputation at the transfemoral level
* Existing prosthesis wearer
* K2/K3/K4 level ambulation
* 18-70 years old
* Mini-Mental State Exam (MMSE) score greater than 17
* Ability to demonstrate proper safety with passive prosthesis
* Candidate for a myoelectric prosthesis (can generate mV level electromyographic EMG signals as detected by surface electrodes
* Candidate for OI surgery as verified by surgical team or has previously received OI
* Candidate for TMR surgery as verified by surgical team or has previously received TMR

Exclusion Criteria:

* Unable to successfully receive osseointegration and TMR
* Significant new injury that would prevent use of a prosthesis: Ability to consistently wear prosthesis and perform activities of daily living and specific performance tasks is necessary to properly evaluate the relative benefits of the intervention
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data.
* Visually impaired
* Proximal nerve injury that prevents TMR
* Individuals who smoke: may interfere with OI process from both bone healing and soft tissue standpoints
* Individuals with active implants.
* Significant comorbidity that would preclude completion of the study, use of prostheses, or would otherwise prevent data acquisition by researchers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Amputee Mobility Predictor with Prosthesis (AMPPRO) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  A questionnaire that measures the ambulatory potential of lower limb amputees. It requires the amputee to complete various tasks. Including sitting balance, reaching, transfers, sit to stand, and standing balance.
Amputee Mobility Predictor with Prosthesis (AMPPRO) | Completion of study, an average of 1 year from enrollment
  A questionnaire that measures the ambulatory potential of lower limb amputees. It requires the amputee to complete various tasks. Including sitting balance, reaching, transfers, sit to stand, and standing balance.
Six Minute Walk Test (6MWT) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The 6 minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Six Minute Walk Test (6MWT) | Completion of study, an average of 1 year from enrollment
  The 6 minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Timed Up and Go (TUG) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults.
Timed Up and Go (TUG) | Completion of study, an average of 1 year from enrollment
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults.
Single Leg Stance Test (SLS) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The Single Leg Stance (SLS) Test is used to assess static postural and balance control. The SLS Test is a balance assessment that is widely used in clinical settings to monitor neurological and musculoskeletal conditions.
Single Leg Stance Test (SLS) | Completion of study, an average of 1 year from enrollment
  The Single Leg Stance (SLS) Test is used to assess static postural and balance control. The SLS Test is a balance assessment that is widely used in clinical settings to monitor neurological and musculoskeletal conditions.
Berg Balance Scale (BBS) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Berg Balance Scale (BBS) | Completion of study, an average of 1 year from enrollment
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Four Square Step Test (FSST) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The Four Square Step Test (FSST) is used to assess dynamic stability and co-ordination. It looks at the ability of the subject to step over low objects forward, sideways, and backward.[
Four Square Step Test (FSST) | Completion of study, an average of 1 year from enrollment
  The Four Square Step Test (FSST) is used to assess dynamic stability and co-ordination. It looks at the ability of the subject to step over low objects forward, sideways, and backward.[
Prosthetic Limb Users Survey of Mobility (PLUS-M) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The Prosthetic Limb Users Survey of Mobility™ is a self-report instrument for measuring mobility of adults with lower limb amputation.
Prosthetic Limb Users Survey of Mobility (PLUS-M) | Completion of study, an average of 1 year from enrollment
  The Prosthetic Limb Users Survey of Mobility™ is a self-report instrument for measuring mobility of adults with lower limb amputation.
Prosthesis Evaluation Questionnaire (PEQ) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The PEQ is a self-evaluating instrument consisting of nine validated scales: ambulation, appearance, frustration, perceived response, stump health, social burden, noise, utility, and well-being.
Prosthesis Evaluation Questionnaire (PEQ) | Completion of study, an average of 1 year from enrollment
  The PEQ is a self-evaluating instrument consisting of nine validated scales: ambulation, appearance, frustration, perceived response, stump health, social burden, noise, utility, and well-being.
Patient Reported Outcome Measure Information System (PROMIS) | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  The PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions.
Patient Reported Outcome Measure Information System (PROMIS) | Completion of study, an average of 1 year from enrollment
  The PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions.

SECONDARY OUTCOMES:
Determine changes in EMG signal quality and neural information resulting from OI and TMR as compared to an instrumented socket for control of a powered leg prosthesis. | Completion of Aim 1:approximately 10-12 weeks (10 in lab visits) from enrollment
  A non-weight bearing independent control system will be configured. The participant will be instructed to attempt to move their 'phantom' limb through knee flexion/extension and ankle plantarflexion/dorsiflexion range movements while EMG data are collected. These data are used to train a pattern recognition control system which can control the leg knee and ankle joints respectively, either in a virtual environment or with the physical prosthesis
Determine changes in EMG signal quality and neural information resulting from OI and TMR as compared to an instrumented socket for control of a powered leg prosthesis. | Completion of study, an average of 1 year from enrollment
  A non-weight bearing independent control system will be configured. The participant will be instructed to attempt to move their 'phantom' limb through knee flexion/extension and ankle plantarflexion/dorsiflexion range movements while EMG data are collected. These data are used to train a pattern recognition control system which can control the leg knee and ankle joints respectively, either in a virtual environment or with the physical prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Levi Hargrove, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No